CLINICAL TRIAL: NCT00645970
Title: Pain, Psychiatric Disorders, and Disability Among Veterans With and Without Polytrauma
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: SDR 07-047
Record Dates: First submitted 2008-03-24; First posted 2008-03-28 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Pain
Keywords: chronic pain; combat injuries; pain assessment; multiple traumas; rehabilitation
MeSH Terms: conditions — Chronic Pain; Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
We believe information to be obtained from this proposed study will prove critical for planning future VA healthcare strategies and developing effective and efficient treatments targeting pain and emotional adjustment difficulties among individuals with polytrauma and returning Operation Enduring Freedom (OEF) and Operation Iraqi Freedom (OIF) personnel. More specifically, this study will be the first to provide systematic data regarding pain and emotional problem prevalence, course, associated impairments, risk factors, and barriers to care and community reintegration among returning OEF and OIF service members with and without polytrauma.

DETAILED DESCRIPTION:
Design Overview: This clinically-oriented study will utilize an observational cohort design to compare cross sectional baseline samples of polytrauma and non-polytrauma OEF/OIF military personnel from two sites (Minneapolis and Tampa VAs) over three time points (baseline and 6 and 12 months post-enrollment). With the relatively large sample sizes employed in this study, cross sectional baseline sampling of existing patients and a longitudinal design will allow us to evaluate associations between injury time and the onset of pain and emotional distress symptoms. The employment of two of the four existing PRCs as study sites will facilitate recruitment of sufficient study participants and will enhance the generalizability of the results. The multiple time points allow us to track the course of pain, emotional problems, and associated disabilities over a 12-month period, and to identify the onset of any new pain or emotional symptoms in participants during the 12-month monitoring period. Most of the study procedures and measures have been utilized in our prior clinical and research efforts with these patient populations. Subjects and Sampling Strategy: Two non-stratified samples of participants will be recruited at each study site. A polytrauma injury group (PTR) will be comprised of between 150 and 200 inpatients or former inpatients returning for additional rehabilitation care to the Minneapolis and Tampa PRCs (ns = 75-100 at each site). PTR subjects will be subdivided into those with combat polytrauma ( 60% based on current data) and those with non-combat polytrauma ( 40%) for selected subsequent analyses. A comparison group of between 300 and 400 non-polytrauma OEF/OIF service members (NPTR) will be sampled randomly from the pool of all veterans on the Minneapolis and Tampa OEF/OIF patient registries (ns = 150-200 at each site). This latter group will be dichotomized into those with pain (NPTR-P; approximately 42 - 50% based on our previous research) and those without (NPTR-NP) for later analyses. Sample Size Determination: The above sample sizes were based on analyses powered to detect significant ( .05) differences in the proportions of pain and PTSD present in the sample cohorts at baseline (H1). For pain, using estimates of pain disorder prevalence among polytrauma (80%) and non-polytrauma (46%) service members based on pain complaint frequencies found in our prior studies,1, 34 and group sizes of 150 (polytrauma) and 300 (non-polytrauma), associated power would approach 1.0. For PTSD, utilizing the same sample sizes and prior research-based estimates of PTSD prevalence rates of 48% (polytrauma) and 32% (non-polytrauma), power to detect a difference between the groups would approach .91. If time allows, we will recruit up to a maximum of 200 PTR and 400 NPTR participants to counter any reduced power due to attrition during the 12-month follow up, to increase the precision of our estimates of the12-month incidence of pain and emotional symptoms in previously symptom-free individuals, and to retain adequate power for subgroup analyses. Inclusionary Criteria - a) PTR group. To participate in the study, PTR subjects must: 1) have been deployed to Iraq or Afghanistan between October 2001 and the present; 2) meet the VA definition of polytrauma injury; 3) receive medical clearance to participate from their attending physician; 4) be able to provide a valid self-report of pain level using the 0-10 Numeric Rating Scale; 5) fluency in verbal and written English; 6) attain a Rancho Los Amigos 35(a scale of cognitive impairment routinely used in PRCs) level of 6 (moderate impairment) or greater; and 7) be competent to provide full informed consent.

Individuals who do not attain Rancho levels exceeding 5 during treatment will not be eligible for participation as in our experience they will be incapable of providing full informed consent or reliable pain scores and will be unable to complete the study self report measures. These criteria were selected to maximize generalizability while minimizing the probability of including polytrauma participants unable to provide valid self-report data. Based on our prior work in this area,1, 34 approximately 70% of PRC patients will attain Rancho levels of 6 or greater and be able to provide valid pain scores during treatment.

Participants may be enrolled at any point during their treatment provided they meet the above criteria. The rationale for allowing enrollment throughout treatment stems from some of the special characteristics of the PTR group. More specifically, polytrauma inpatients often are admitted on large doses of opioid analgesics which may limit their ability to provide reliable self-reports of pain, particularly if they also have experienced a TBI. As the opioid dosages are titrated in order to promote increased involvement in rehabilitation, they may be more able to provide valid pain ratings. Secondly, the cognitive function of soldiers with significant cognitive limitations typically improves substantially during treatment,1, 34 sometimes dramatically. If we were to limit participation only to those able to provide valid self-reports of pain or other symptoms at the time of admission we would restrict the pool of potential participants and substantially reduce the generalizability and clinical utility of the study. Because we are not focusing on treatment effects, and because we are using a cross-sectional baseline sampling approach and will be controlling for time since injury, this approach will not bias the obtained data. b) NPTR group. Criteria for NPTR participation include: 1) deployment to Iraq or Afghanistan between October 2001 and the present; 2) fluency in verbal and written English; 3) ability to provide a valid self-report of pain level using the 0-10 Numeric Rating Scale; and 4) competency to give full informed consent. This comparison group will include participants who do not meet polytrauma criteria and be sampled from all eligible members of the registries of both participating VA facilities. Participants who meet the above criteria will be enrolled for one-year. Women and minorities will be recruited to the extent that they are present in the associated participant pools, but will not be oversampled. Participants will receive a token payment of $30 following each completed assessment session in order to defray their travel expenses and time investments. Estimated Participation Rates and Participant Pool Size. Based on our experience in recruiting participants for prior chronic pain, polytrauma, and OEF/OIF studies or clinical evaluations, we anticipate that at least 80% of those who meet the study criteria will agree to participate. Therefore, in order to meet our minimum recruitment goals we will need at least 280 individuals with polytrauma (280 X 67% able to provide pain ratings X 80% participation rate = 150). In the past 12 months, a total of 490 individuals have been admitted or returned to the Minneapolis (n=289) and Tampa (n=201) PRCs, suggesting a more than adequate pool of participants with polytrauma. Minimum recruitment goals for OEF/OIF soldiers without polytrauma will require a participant pool of at least 376 individuals (376 X 80% participation rate = 300). As of May 1st, 2007, there are 3723 OEF/PIF returnees on the Minneapolis OEF/OIF registry, and 4099 on the Tampa patient registry.

ELIGIBILITY:
Inclusion Criteria:

for Polytrauma Participants

* Was deployed to Iraq or Afghanistan between October 2001 and the present
* Meets the VA definition of polytrauma injury
* Received medical clearance from attending physician to participate in study
* Able to provide valid self-report of pain level using 0-10 numeric rating scale
* Fluent in verbal and written English
* Rancho Los Amigos level 6
* Competent to provide full informed consent

for Non-Polytrauma Participants

* Was deployed to Iraq or Afghanistan between October 2001 and the present
* Fluent in verbal and written English
* Able to provide valid self-report of pain level using 0-10 numeric rating scale
* Competent to provide full informed consent

Exclusion Criteria:

see above.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Two non-stratified samples of participants will be recruited at each study site. A polytrauma injury group (PTR) will be comprised of between 150 and 200 inpatients or former inpatients returning for additional rehabilitation care to the Minneapolis and Tampa PRCs (ns = 75-100 at each site). PTR subjects will be subdivided into those with combat polytrauma (60% based on current data) and those with non-combat polytrauma (40%) for selected subsequent analyses. A comparison group of between 300 and 400 non-polytrauma OEF/OIF service members (NPTR) will be sampled randomly from the pool of all veterans on the Minneapolis and Tampa OEF/OIF patient registries (ns = 150-200 at each site). This latter group will be dichotomized into those with pain (NPTR-P; approximately 42 - 50% based on our previous research) and those without (NPTR-NP) for later analyses.
Sampling Method: Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2008-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Clark, PhD MA, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (1):
- James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida, United States

REFERENCES:
- [Background] Buckenmaier III CC, Gallagher RM, Cahana A, Clark ME, Davis SA, Brandon-Edwards H, Griffith S, Houston JS, Jankovich E, Kurihara C, Mackey S, Rupprecht C, Spevak C. War on Pain: New Strategies in Pain Management for Military Personnel and Veterans. Federal practitioner : for the health care professionals of the VA, DoD, and PHS. 2011 Jan 1; 28(Suppl 2):1-16.
- [Background] Kalra R, Clark ME, Scholten JD, Murphy JL, Clements KL. Managing pain among returning service members. Federal practitioner : for the health care professionals of the VA, DoD, and PHS. 2008 Jan 1; 25:36-45.
- [Result] Lew HL, Otis JD, Tun C, Kerns RD, Clark ME, Cifu DX. Prevalence of chronic pain, posttraumatic stress disorder, and persistent postconcussive symptoms in OIF/OEF veterans: polytrauma clinical triad. J Rehabil Res Dev. 2009;46(6):697-702. doi: 10.1682/jrrd.2009.01.0006. PMID 20104399
- [Result] Walker RL, Clark ME, Nampiaparampil DE, McIlvried L, Gold MS, Okonkwo R, Kerns RD. The hazards of war: blast injury headache. J Pain. 2010 Apr;11(4):297-302. doi: 10.1016/j.jpain.2009.12.001. No abstract available. PMID 20350705
- [Result] Dobscha SK, Clark ME, Morasco BJ, Freeman M, Campbell R, Helfand M. Systematic review of the literature on pain in patients with polytrauma including traumatic brain injury. Pain Med. 2009 Oct;10(7):1200-17. doi: 10.1111/j.1526-4637.2009.00721.x. PMID 19818031
- [Result] Gironda RJ, Clark ME, Ruff RL, Chait S, Craine M, Walker R, Scholten J. Traumatic brain injury, polytrauma, and pain: challenges and treatment strategies for the polytrauma rehabilitation. Rehabil Psychol. 2009 Aug;54(3):247-58. doi: 10.1037/a0016906. PMID 19702423
- [Result] Clark ME. Cost-effectiveness of multidisciplinary pain treatment: are we there yet? Pain Med. 2009 Jul-Aug;10(5):778-9. doi: 10.1111/j.1526-4637.2009.00659.x. No abstract available. PMID 19691153
- [Result] Clark ME, Scholten JD, Walker RL, Gironda RJ. Assessment and treatment of pain associated with combat-related polytrauma. Pain Med. 2009 Apr;10(3):456-69. doi: 10.1111/j.1526-4637.2009.00589.x. PMID 19416437
- [Result] Clark ME, Walker RL, Gironda RJ, Scholten JD. Comparison of pain and emotional symptoms in soldiers with polytrauma: unique aspects of blast exposure. Pain Med. 2009 Apr;10(3):447-55. doi: 10.1111/j.1526-4637.2009.00590.x. PMID 19416436
- [Result] Clark ME, Hooten WM, Sanders SH. Interdisciplinary pain rehabilitation: current challenges and future opportunities. Pain Med. 2011 Jan;12(1):152-3. doi: 10.1111/j.1526-4637.2010.01034.x. No abstract available. PMID 21223493
- [Result] Walker RL, Clark ME, Sanders SH. The Postdeployment multi-symptom disorder: An emerging syndrome in need of a new treatment paradigm. Psychological Services. 2010 Aug 1; 7(3):136-147.

RESULTS

PARTICIPANT FLOW:
Groups:
- Polytrauma System of Care (PSC): Participants recruited from the Polytrauma System of Care (PSC)
- Registry: Participants recruited from the OEF/OIF/OND registry
Period: Overall Study
Arm/Group | Polytrauma System of Care (PSC) | Registry
Started | 141 | 218
6 Months | 58 | 97
1 Year | 37 | 42
Completed | 32 | 32
Not Completed | 109 | 186

BASELINE CHARACTERISTICS:
Groups:
- Polytrauma System of Care (PSC): Participants recruited from the Polytrauma System of Care
- Total: Total of all reporting groups
Arm/Group | Polytrauma System of Care (PSC) | Registry | Total
Number analyzed (Participants) | 141 | 218 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (8.2) | 36.6 (10.3) | 35.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 22 | 32
  Male | 131 | 196 | 327
Race/Ethnicity, Customized [Number; unit: participants]
  White | 120 | 158 | 278
  Hispanic | 13 | 23 | 36
  Black | 7 | 27 | 34
  Other | 1 | 10 | 11

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scales of Pain Over Past Week (11 Point Likert Scale)
Description: Numeric Pain Rating Scale is a self-report measure of "usual" (average) pain intensity over the last week; response options range from "no pain" (0) to "worst pain imaginable" (10). A score >3 indicates moderate-to-severe pain.
Time Frame: Baseline, 6 months, 1 year
Population: Numeric Pain Rating Scale data are missing for 21 participants (PSC n=1; Registry n=20)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Polytrauma System of Care (PSC) | Registry
Number analyzed (Participants) | 140 | 198
units on a scale
  Baseline | 4.66 (2.44) | 3.80 (2.46)
  6 months | 4.92 (2.20) | 3.30 (2.36)
  1 year | 4.88 (3.02) | 4.69 (2.89)

ADVERSE EVENTS:
Arm/Group | Polytrauma System of Care (PSC) | Registry
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/218
Other Adverse Events (participants affected / at risk) | 0/141 | 0/218

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No